CLINICAL TRIAL: NCT05050448
Title: Comparative Usability Evaluation of Sustained Acoustic Medicine (SAM) Devices and Topical Gel for Knee Pain Related to Osteoarthritis
Brief Title: Comparative Usability Evaluation of Sustained Acoustic Medicine (SAM) Devices and Topical Gel for OA Knee Pain
Status: Completed | Phase: Phase 1 / Phase 2 | Type: Interventional
Sponsor: ZetrOZ, Inc. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: HF-01-2021
Record Dates: First submitted 2021-09-09; First posted 2021-09-20 (Actual); Results first posted 2025-05-02 (Actual); Last update posted 2025-05-02 (Actual); Status verified 2025-04

CONDITIONS: Knee Osteoarthritis
Keywords: Non-Steroidal Anti-Inflammatory Drugs; Sustained Acoustic Medication; Low-Intensity Continuous Ultrasound
MeSH Terms: conditions — Osteoarthritis, Knee | interventions — Diclofenac

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: Yes

ARMS (3):
- SAM Ultrasound Device and Diclofenac Patch (Experimental): Patients receive treatment from the wired SAM Ultrasonic Diathermy Device for 4 hours at least 5 days a week for 8 weeks combined with 2.5% diclofenac patch. The SAM device emits continuous ultrasound at 3 megahertz (MHz) frequency and 0.132 watts/cm2 intensity.
  Interventions: Device: Sustained Acoustic Device with 2.5% Diclofenac Patch
- SAM2 Ultrasound Device and Diclofenac Patch (Experimental): Patients receive treatment from the wireless SAM Ultrasonic Diathermy Device for 1 hour at least 5 days a week for 8 weeks combined with 2.5% diclofenac patch. The SAM device emits continuous ultrasound at 3 megahertz (MHz) frequency and 0.132 watts/cm2 intensity.
  Interventions: Device: Sustained Acoustic Device with 2.5% Diclofenac Patch
- Topical Pain-Relief Gel (Placebo Comparator): Patients apply topical 1% diclofenac gel three times per day, at least 5 days per week for 8 weeks.
  Interventions: Drug: 1% Diclofenac Topical Gel

INTERVENTIONS:
Device: Sustained Acoustic Device with 2.5% Diclofenac Patch — Patients apply the SAM Ultrasonic Diathermy Device daily for 1-4 hours of continuous therapeutic ultrasound at 3 megahertz(MHz) frequency and 0.132 Watts/cm@ with 2.5% Diclofenac patches.
  Other Names: ZetrOZ Ultrasound Device; Wearable Ultrasound Device; Long Duration Ultrasound; LITUS Device; Long Duration Low-Intensity Device
  Arms: SAM Ultrasound Device and Diclofenac Patch; SAM2 Ultrasound Device and Diclofenac Patch
Drug: 1% Diclofenac Topical Gel — Topical pain-relief gel
  Other Names: Voltaren
  Arms: Topical Pain-Relief Gel

SUMMARY:
The purpose of this study is to evaluate the usability of the ultrasound devices and common pain relief gel. The ability of the three treatment approaches to reduce pain, stiffness, and functionality as measured by NRS scale and the Western Ontario and McMaster Universities Arthritis Index (WOMAC) will be evaluated.

ELIGIBILITY:
Inclusion Criteria:

* Physician-diagnosed mild to moderate knee osteoarthritis (KL Grade 2-3) based on fixed-flexion x-ray radiological findings for osteophytes and joint space narrowing within the past 12 months
* Fulfill the American College of Rheumatology clinical and radiological diagnostic criteria for knee OA
* 35-80 years of age
* Report a frequent pain score between 4-7 (NRS range: 0-10) during the week preceding enrollment
* Report that knee pain negatively affects quality of life
* Willing not to use any cream, gel, or topical solution during the administration of treatment other than the approved ultrasound gel provided to the subject at the initiation of the study
* Deemed appropriate by their physician or by the study site physician to participate
* Willing and able to self-administer treatment daily within their place of residence or during normal daily activity, excluding bathing, showering, or other water activities which may result in submersion of the study device
* Not initiate use of opioid and/or non-opioid analgesic medications
* Willing to discontinue any other interventional treatment modalities on the knee during the study period

Exclusion Criteria:

* Cannot successfully demonstrate the ability to put on and take off the device
* Display any condition which, in the judgment of the investigator, would make participation in the study unacceptable, including, but not limited to, the subject's ability to understand and follow instructions
* Have severe OA or have little to no cartilage in the knee
* Have knee replacement, other surgical intervention, or hyaluronidase injection in the affected knee in the past 6 months
* Is non-ambulatory (unable to walk)
* Is pregnant
* Is a prisoner
* Has a pacemaker
* Has a malignancy in the treatment area
* Has an active infection, open sores, or wounds in the treatment area
* Has impaired sensation in the treatment area, such as caused by chemotherapy or anesthesia
* Has known neuropathy
* Has a hereditary disposition (tendency) for excessive bleeding (hemorrhage)
* Participated in a clinical trial for an investigational drug and/or agent within 30 days prior to screening
* Modify their medications during the course of the study (medications and doses must remain constant throughout the study)
* Currently taking steroids
* Have contraindication to radiograph
* Have a secondary cause of arthritis (metabolic or inflammatory)

Ages: 35 Years to 80 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 60 (Actual)
Dates: Start 2021-08-01 (Actual); Primary Completion 2022-12-01 (Actual); Study Completion 2022-12-31 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: George K Lewis, Ph.D., Principal Investigator — ZetrOZ Systems
Locations (3):
- United States (3):
  - Orthopaedic Foundation, Stamford, Connecticut
  - ZetrOZ Systems, Trumbull, Connecticut
  - Cayuga Medical Center - Medical Pain Consultants, Dryden, New York

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- See also: Class II Medical Device — https://www.samrecover.com

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | SAM Ultrasound Device and Diclofenac Patch | SAM2 Ultrasound Device and Diclofenac Patch | Topical Pain-Relief Gel
Started | 20 | 20 | 20
Completed | 17 | 17 | 18
Not Completed | 3 | 3 | 2

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | SAM Ultrasound Device and Diclofenac Patch | SAM2 Ultrasound Device and Diclofenac Patch | Topical Pain-Relief Gel | Total
Number analyzed (Participants) | 20 | 20 | 20 | 60
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0 | 0 | 0 | 0
  Between 18 and 65 years | 20 | 20 | 20 | 60
  >=65 years | 0 | 0 | 0 | 0
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 10 | 10 | 10 | 30
  Male | 10 | 10 | 10 | 30
Race and Ethnicity Not Collected [Count of Participants; unit: Participants] — Population: Race and Ethnicity were not collected from any participant.

OUTCOME MEASURES:

1. Primary Outcome: Change in Pain Units on a Scale (0-10) 0 Being Least, 10 Being Worst Pain From Baseline
Description: Change in the self described pain units on a scale by patient at baseline and post-treatment on the range of 0 - 10, 0 being the least pain and 10 being the worst pain.
Time Frame: 8 weeks
Measure: Mean (Standard Error); unit: units on a scale
Arm/Group | SAM Ultrasound Device and Diclofenac Patch | SAM2 Ultrasound Device and Diclofenac Patch | Topical Pain-Relief Gel
Number analyzed (Participants) | 17 | 17 | 18
units on a scale | -3.56 (0.37) | -3.29 (0.41) | -1.00 (0.37)

2. Primary Outcome: Change in the Western Ontario and McMaster Universities Osteoarthritis Index (WOMAC) From Baseline
Description: WOMAC questionnaire will be utilized (Western Ontario and McMaster Universities Arthritis Index) at baseline and post-treatment to calculate the change in scores. Total score is the sum of pain, stiffness, and function scores (range of 0 - 96). A higher score is considered a worse outcome, and a lower score is considered a better outcome.
Time Frame: 8 weeks
Measure: Mean (Standard Error); unit: units on a scale
Arm/Group | SAM Ultrasound Device and Diclofenac Patch | SAM2 Ultrasound Device and Diclofenac Patch | Topical Pain-Relief Gel
Number analyzed (Participants) | 17 | 17 | 18
units on a scale | -15.71 (2.31) | -16.71 (4.87) | -5.72 (2.31)

ADVERSE EVENTS:
Time Frame: 1 year
Arm/Group | SAM Ultrasound Device and Diclofenac Patch | SAM2 Ultrasound Device and Diclofenac Patch | Topical Pain-Relief Gel
All-Cause Mortality (participants affected / at risk) | 0/20 | 0/20 | 0/20
Serious Adverse Events (participants affected / at risk) | 0/20 | 0/20 | 0/20
Other Adverse Events (participants affected / at risk) | 0/20 | 0/20 | 0/20

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2021-05-20): https://cdn.clinicaltrials.gov/large-docs/48/NCT05050448/Prot_SAP_002.pdf